CLINICAL TRIAL: NCT01322503
Title: Evaluation of the Susceptibility of Human Volunteers With Different Histo-Blood Group Antigens to Norovirus
Brief Title: Susceptibility of Human Volunteers With Different Histo-Blood With Different Histo-Blood Group Antigens to Norovirus
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Quadruple
Other Study IDs: PR033018
Record Dates: First submitted 2010-10-25; First posted 2011-03-24 (Estimated); Last update posted 2012-02-10 (Estimated); Status verified 2012-02

CONDITIONS: Healthy Adults

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Norovirus Challenge (Experimental)
  Interventions: Biological: Norovirus
- Norovirus challenge (Experimental)
  Interventions: Biological: Norovirus

INTERVENTIONS:
Biological: Norovirus — Norovirus challenge pool administered to each subject
  Other Names: Norovirus challenge pool

SUMMARY:
Objectives: To evaluate the role of human histo-blood group antigens in susceptibility to Norovirus infections.

Description of Study Design: Healthy volunteers with different blood types and low antibody titers to the challenge strain will be challenged orally with a Norovirus in the CCCR inpatient facility. Subjects with resistant (non-secretors) or susceptible (secretors (of either A, B or O blood group)) to the challenge strain will be recruited. The challenge study will be conducted in two groups of twenty, each with approximately ten secretors and ten non-secretors. Three additional subjects per group will serve as alternates in the event that any of the study subjects are unavailable or become ineligible at the time of the inpatient study. Subjects will be monitored daily in the isolation facility for at least five days following this challenge for daily clinical and virological evaluations. Subjects will return to the investigational site for evaluation the day after discharge from the inpatient unit and about 30 days (28-35 days) post challenge.

Study Endpoints: Norovirus infection as assessed by viral shedding, seroconversion and clinical illness assessed by the duration and severity of symptoms

DETAILED DESCRIPTION:
Noroviruses are single-stranded, positive-sense RNA viruses that cause acute gastroenteritis in humans. The prototype Norwalk virus (NV) was identified in a large outbreak of acute gastroenteritis in an elementary school in Norwalk, Ohio, in 1968. Since then, many strains have been described and named by the locations of their first isolation. Genetically, Noroviruses belong to one of four genera within Caliciviridae (CV). Phylogenetic analysis has shown that the Norovirus genus is divided into five genogroups and each genogroup can be further divided into genetic clusters; at least 30 genetic clusters of Noroviruses have been identified.

Noroviruses have been recognized as the most important cause of non-bacterial epidemics of acute gastroenteritis, affecting individuals of all ages, in both developing and developed countries. Such outbreaks usually have high attack rates and have occurred in child care centers, schools, restaurants, summer camps, hospitals, nursing homes, ships (both civilian and military) as well as deployed military troops. The viruses are highly contagious and are able to survive in the environment for extended periods of time. They are spread by contact with environmental surfaces and person-to-person transmission. Noroviruses normally cause moderate-to-severe diarrhea and the disease is often incapacitating and can be fatal in the young and elderly. The most important public health concern is that Noroviruses can cause large water- and food-borne outbreaks, resulting in the virus being classified as a Category B agent.

Noroviruses have also been implicated in several military outbreaks. The "Desert Shield virus" (DSV) isolated in US troops in the 1991 Gulf War was subsequently identified as a Norovirus. Similarly the recently reported "mysterious" attacks of acute gastroenteritis affecting the British troops in Afghanistan were also caused by a Norovirus. Large outbreaks of Norovirus-associated gastroenteritis are common on US Navy ships, similar to those that occurred on board cruise ship lines. Surveillance of acute gastroenteritis on board five US Navy combat ships in 1998-1999 showed that all the ships experienced large outbreaks of Norovirus acute gastroenteritis during their deployment in the Pacific and Indian Oceans, following port visits. Because of the rapid spread of the disease, many departments and units on board the ships were unable to function during the peak of the outbreaks.

Noroviruses are difficult to study because: 1) they are genetically and antigenically highly diverse and multiple strains with distinct genetic identities co-circulate in the same communities, making diagnosis and disease control extremely difficult; and 2) the virus cannot be cultivated in cell culture and 3) no small animal model for studying Noroviruses exists. The molecular cloning of the prototype Norwalk Virus (NV) in 1990 by one of the co-investigators of this application has allowed rapid progress in studying Noroviruses and other genera; however, many issues on Norovirus infection, pathogenesis, immunology and host range remain unknown.

The discovery of Norovirus receptors provides new opportunities to evaluate the pathogenesis and epidemiology of Noroviruses. A host genetic factor involving Norovirus infection was originally suggested by many researchers before the cloning of Noroviruses in the 1990s because about 20-30% of individuals who did not have antibodies against Noroviruses were never infected following a challenge with NV, and in outbreaks, individuals who remained healthy were clustered in families that had the same exposure to Noroviruses as the ill families. Further, pre-existing antibodies against NV were not protective against NV infection, while individuals who had high levels of antibodies against NV were more susceptible to NV than individuals who did not have the antibodies. These observations indicate that, in addition to immune responses, there must be another factor(s) that controls the host-specificity of Norovirus infection.

We recently discovered that Noroviruses recognize human histo-blood group antigens as receptors. Using recombinant capsid proteins from different Noroviruses representing different genetic clusters, we have identified four binding patterns of Noroviruses to human histo-blood group antigens, which are defined by the host Lewis, secretor and ABO blood types. This finding provides a new approach to develop strategies to control the disease. Specifically, if Noroviruses rely on the histo-blood group antigens on the surfaces of the intestinal epithelial cells as receptors, a compound that inhibits the interaction between the virus and receptors could be developed as an antiviral drug for Noroviruses. This finding provides the basis for this protocol which seeks to confirm the relationship between specific Norovirus susceptibility and specific histo-blood group antigen presence as well as establish a model to evaluated future interventions (drugs and vaccines).

The specificity of the NV interaction with the sugar moieties of histo-blood group antigens was shown by specific blocking of the binding by human milk from a secretor, by monoclonal antibodies specific for secretor human blood-group antigens (HBGAs), by synthetic oligosaccharide conjugates containing secretor antigens, and by treatment of the tissues with a1,2 fucosidase. NV also binds to differentiated CaCo2 cells and differentiated CaCo2 cells express human histo-blood group antigens. Transfection of Chinese Hamster Ovary (CHO) cells with a a1,2-linked fucosyl-transferase cDNA allowed attachment of NV virus-like particles (VLPs). The bound rNV VLPs were internalized following incubation of the cells at 37oC.

To further investigate the association between secretor status and susceptibility to Norwalk virus (NV), we collaborated with Dr. Christine Moe at Emory University's School of Medicine on a volunteer challenge study. This study utilized the prototype NV, the first Norovirus strain to be used for human challenge studies. Saliva samples from 77 NV-challenged volunteers were tested for secretor status and for NV-binding. Fifty-five (71%) of the 77 volunteers were secretors. Among the 55 secretors, 34 (62%) were infected with NV following challenge and saliva from 41 (75%) bound NV recombinant VLPs. None of the saliva samples from the 22 non-secretor volunteers bound NV virus-like particles (VLPs) and none of them became infected following NV challenge; strongly suggesting that the susceptibility to NV is determined at least in part by the ability of the host to bind the norovirus strain.

More recently we performed a study to determine whether other strains of Noroviruses have a similar pattern of host-specificity and have extended the binding patterns to 7 based on examination of fourteen Noroviruses. The 7 patterns have been classified into two groups according to their interactions with three major epitopes (A/B, H and Lewis) of HBGAs: the A/B binding group and the Lewis-binding group. Strains in the A/B binding group recognize the A and/or B and H antigens, but not the Lewis antigens, while strains in the Lewis-binding group react only to the Lewis and/or H antigens. This classification also resulted in a model of the Norovirus/HBGA interaction, in which a maximum of two binding sites within a receptor binding interface are involved in NV/HBGA interaction. The A, B and H side chains are responsible for binding by the A/B binding strains while the Lewis epitopes are responsible for the Lewis binding strains. Phylogenetic analyses showed that strains with identical or closely related binding patterns tended to be clustered, but strains in both binding groups can be found in both genogroups I and II. Our results suggest that Noroviruses have a wide spectrum of host range and human HBGAs play an important role in Norovirus evolution.

Since human Noroviruses cannot be cultivated in vitro or infect animals, it is necessary to perform human volunteer challenge studies to study the pathobiology of the infection. The study will further the concept that Norovirus has a narrow host range which is fundamental in the pathogenesis and immunology of Noroviruses. Additionally, we recently have identified more than a dozen compounds that specifically block Norovirus attachment to their receptors. The human challenge study should also establish a model that can be used in the evaluation of these new compounds in regards to their capacity to block virus replication (anti-viral drug). Furthermore, our study will re-evaluate whether acquired immunity is an independent factor in Norovirus infections which may provide additional information in host immunity potentially useful in vaccine development. Finally, the study will allow for banking of the Norovirus challenge strain by collecting the diarrheal stools passed by the study subjects. Banking of additional specimen, as mentioned above, is critical for future clinical trials because the virus cannot be cultivated in vitro and must be isolated from humans infected with the virus.

A specific challenge study would only use one challenge strain and any challenge strain used in human clinical trials would have a separate IND and FDA approval prior to administration to subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults between the ages of 18 and 49 years
* Willing and able to provide written informed consent
* Able to comply with all study procedures
* Have a body mass index of at least 19
* Have a serum IgG antibody titer of < 1:1,600 to Norovirus
* Female subjects of child bearing potential must have negative urine pregnancy tests
* Female subjects must be of non-childbearing potential, or if of childbearing potential (as determined by investigator) must be practicing abstinence or using an effective licensed method of birth control for one month before receipt of challenge through one month after completing the inpatient isolation facility stay.
* Have normal screening laboratories
* Score at least 70% on a test of understanding of this research study.

Exclusion Criteria:

* Expected to be noncompliant with study procedures or planning to move within the anticipated total duration of the study
* Pregnant or breastfeeding
* HIV, Hepatitis B or C positive
* Norovirus antibody screening titer of > 1:1600
* Clinically significant findings on history or physical examination
* Clinically significant history of diseases or treatments that may affect the immune system's function
* Receipt of systemic corticosteroids for greater than 7 days within the past six months
* Abnormal screening electrocardiogram (ECG)
* Clinically significant respiratory disease, endocrine disease, liver disease, renal disease, or neurological disease
* History of malabsorption or maldigestion disorder, major gastrointestinal (GI) surgery, or any other chronic GI disorders that would interfere with the study
* Clinically significant abnormalities of the health screening laboratory work
* Use of antibiotics within 7 days prior to entry into the inpatient isolation facility (Day -1)
* Any medical illness requiring a new prescription medication or hospitalization during the screening period
* Temperature ≥38.0°C
* Diarrhea or vomiting during the 7 days prior to challenge administration
* Allergy to sodium bicarbonate solution
* Treatment within the past year for an eating disorder
* History of alcohol or drug abuse within past 3 years
* Receipt of any vaccine, licensed or investigational, or any investigational product within 30 days of challenge administration or plan to receive any vaccine or investigational product through the study duration
* Use of any H2 receptor antagonists or prescription acid suppression medication or over-the-counter (OTC) antacids within 72 hours of investigational product administration (Day 0)
* Use of prescription and OTC medications containing acetaminophen, aspirin, ibuprofen, and other non-steriodal anti-inflammatory drugs within 48 hours prior to investigational product administration
* Regular use of laxatives or anti-motility agents
* Receipt of blood or blood products within the past six months
* Subjects who are unwilling or unable to cease smoking for the duration of the inpatient stay
* Any other condition, such as a medical, psychiatric, or social condition or occupational responsibility that, in the judgment of the investigator, would interfere with or serve as a contraindication to the subject's participation in the study or assessment of the investigational product
* Plan to be living in a confined environment within 3 weeks after receiving the challenge strain
* Commercial food handlers, day care workers, or health care workers involved in direct patient contact
* Provide child day care services either in a home or in a nonresidential facility
* Provide direct care to individuals over 65 years of age, young children (<2 years) at home or with household contacts who are:

  * Immunocompromised
  * Pregnant, or
  * Breast feeding

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2010-10; Primary Completion 2011-02 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Measurement of the number of people who develop symptomatic illness after challenge with Norovirus | 1 month after challenge
  The number of subjects that become infected, as measured by the number of subjects found to be shedding norovirus in their stool, as well as the number of symptomatic infections (viral shedding in addition to other symptoms such as vomiting, diarrhea, abdominal cramps) will be the primary outcome measure.
  We will also assess the number of subjects who show at least a 4-fold rise in antibodies against Norovirus (comparing pre-challenge and post-challenge antibody levels).

CONTACTS AND LOCATIONS:
Overall Officials: Robert Frenck, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

REFERENCES:
- [Derived] Frenck R, Bernstein DI, Xia M, Huang P, Zhong W, Parker S, Dickey M, McNeal M, Jiang X. Predicting susceptibility to norovirus GII.4 by use of a challenge model involving humans. J Infect Dis. 2012 Nov;206(9):1386-93. doi: 10.1093/infdis/jis514. Epub 2012 Aug 20. PMID 22927452